CLINICAL TRIAL: NCT05527535
Title: Expansion of Integrated AI Solution for Diabetic Retinopathy Screening in Thailand: An Implementation Research
Brief Title: Expansion of Integrated AI Solution for Diabetic Retinopathy Screening in Thailand
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Department of Medical Services Ministry of Public Health of Thailand (Other Government)
Collaborators: Health Systems Research Institute,Thailand (Other Government)
Responsible Party: Sponsor
Other Study IDs: 65057
Record Dates: First submitted 2022-08-25; First posted 2022-09-02 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-08

CONDITIONS: Diabetic Retinopathy
Keywords: Diabetic Retinopathy, Screening, Deep Learning Algorithm, Human Grader
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- AI screening group: Diabetes mellitus patients undergo diabetic retinopathy screening by AI
  Interventions: Diagnostic Test: Diabetic retinopathy screening by artificial intelligence
- Manual screening group: Diabetes mellitus patients undergo diabetic retinopathy screening by health care personnel
  Interventions: Diagnostic Test: Diabetic retinopathy screening by healthcare personnel

INTERVENTIONS:
Diagnostic Test: Diabetic retinopathy screening by artificial intelligence — Screening diabetic patients' eyes with AI through digital health platform
  Groups: AI screening group
Diagnostic Test: Diabetic retinopathy screening by healthcare personnel — Screening diabetic patients' eyes by conventional method (healthcare personnel)
  Groups: Manual screening group

SUMMARY:
Efficiency and effectiveness of real-world diabetic retinopathy screening by artificial intelligent (AI) are limited. Investigators will implement AI for diabetic retinopathy screening in 13 health districts in Thailand and investigate the efficiency, effectiveness as well as patients and health care personnel's satisfaction by an implementation research.

ELIGIBILITY:
Inclusion Criteria:

1. Type 1 or 2 diabetes mellitus patients whose name are in primary hospital record
2. No full-time ophthalmologists in those primary hospital
3. Age more than or equal to 18 years
4. Eligible for fundus photo imaging at least 1 eye

Exclusion Criteria:

1. Type 1 or 2 diabetes mellitus patients whose name are in primary hospital record that have full-time ophthalmologists
2. Patients who previously diagnosed with other causes of macular edema, for example, Age-related Macular Degeneration, Radiation Retinopathy, Retinal Vein Occlusion etc.
3. History of retinal laser or surgery
4. Other ocular diseases that require referral to ophthalmologists
5. Not eligible for fundus photo imaging for both eyes (any causes)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All diabetes mellitus patients who visit for diabetic retinopathy screening at selected primary care units and hospitals in 13 health districts in Thailand
Sampling Method: Non-Probability Sample
Enrollment: 34500 (Estimated)
Dates: Start 2022-10-03 (Estimated); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of AI in diabetic retinopathy screening | Throughout the whole period of screening, approximately 6 months
  Referral adherance of patients in AI group in percentage
Efficiency of AI in diabetic retinopathy screening | Throughout the whole period of screening, approximately 6 months
  Down time and failure rate of AI system
Efficiency of AI in diabetic retinopathy screening | Throughout the whole period of screening, approximately 6 months
  Cost in development and implement of AI system in Thai baht unit

SECONDARY OUTCOMES:
Satisfaction of patients and health care personnel in AI-based screening | At the end of the screening, approximately at Month 6
  Measurement of health care personnel's satisfaction by well-developed questionnaire

IPD SHARING:
Plan to Share IPD: No
Fear of inappropriate use of data